CLINICAL TRIAL: NCT00291512
Title: Promoting Safer Sex in HIV+ MSM Methamphetamine Users
Brief Title: Promoting Safer Sex in HIV+ Homosexual and Bisexual Men Who Use Methamphetamine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DESPR DA012116; R01DA012116 (NIH)
Record Dates: First submitted 2006-02-10; First posted 2006-02-14 (Estimated); Last update posted 2011-10-13 (Estimated); Status verified 2008-11

CONDITIONS: HIV Infections; STDs; Methamphetamine Abuse
Keywords: HIV; STDs; Methamphetamine abuse; MSM
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases

INTERVENTIONS:
Behavioral: Theory-based counseling program

SUMMARY:
This project studies the effectiveness of a sexual risk reduction intervention among HIV+ Men who have Sex with Men (MSM) and who use methamphetamine.

ELIGIBILITY:
Inclusion Criteria:

* HIV+
* Men who have sex with men

Exclusion Criteria:

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L. Patterson, Ph.D., Principal Investigator — University of California, San Diego
Locations (1):
- HIV Neurobehavioral Research Center, San Diego, California, United States